CLINICAL TRIAL: NCT05959876
Title: The Effect of Training on Perineal Care of Palliative Care Patients With Incontinence on the Knowledge Level of Relatives: A Randomized Controlled Study
Brief Title: The Effect of Perineal Care Education on Palliative Care Patient' Relatives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Lutfiye Nur Uzun, PhD Nurse, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-HEM-UZUN-003
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Perineum Care; Caregiver Education; Palliative Care
MeSH Terms: interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study with experimental and control groups consisting of pre-test and post-test
Who Masked: Outcomes Assessor
Masking Description: Outcome evaluations will be conducted by a researcher blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Face-to-face perineal care training will be given to the relatives of the patients in the training group in the determined common time period. During the trainings, the presentation prepared in the power point program and the content of perineum care will be conveyed by the researcher in two 30-minute sessions using plain lecture, case study and question and answer techniques.
  Interventions: Other: Training group
- Control group (Active Comparator): The participants in the control group will not be interfered with by the researcher during the research.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Training group — Face-to-face perineal care training
  Arms: Training group
Other: Control group — No intervention
  Arms: Control group

SUMMARY:
The aim of this randomized controlled study, which includes pre-test and post-test, is to examine the perineum care education given to caregivers of patients with incontinence and being treated in a palliative care clinic.

The basic question it aims to answer is:

Does the perineum care training given to the relatives of patients treated in the palliative care clinic have an effect on the level of knowledge about perineum care?

Participants will participate in a training activity on perineum care. Researchers will compare whether perineum care training given to relatives of palliative care patients is effective compared to the routine service operation, by using lecture, question-answer and presentation method.

DETAILED DESCRIPTION:
A time period suitable for the clinic, patient and companion will be determined by making one-to-one interviews with the companions in the experimental and control groups. Care will be taken to make the applications outside of treatment, visit, care, meal and visitor hours. Accompanying attendants will be met at the specified time and information about the work will be given.

Participants in the control group will be given a Personal Information Form and a Perineum Care Knowledge Test as a pre-test and will be given sufficient time to complete them. The participants in the control group will not be interfered with by the researcher during the research. At the end of the same day, the Perineum Care Knowledge Test will be redistributed and collected as a posttest to the control group. This group will only receive routine nursing training given in the hospital. In palliative care clinics, nurses provide information to patients and their families to help patients maintain their independence and control and make choices during their daily care. In addition, trainings are planned for the needs of the patient and his family. After the research process is completed, a handbook on perineal care will be distributed to the participants in the control group by the researcher.

The participants in the experimental group will be given a Personal Information Form and a Perineum Care Knowledge Test as a pre-test and will be given sufficient time to fill them out. Face-to-face and one-to-one perineal care training will be given to the participants in the experimental group. During the trainings, the presentation prepared in the power point program and the content of perineum care will be conveyed by the researcher in two 30-minute sessions using plain lecture, case study and question and answer techniques. These techniques used are considered to be effective methods in the education of patients and their relatives. Opinions were received from three field experts regarding the content validity of the content of perineal care (CGI: 1.00). The Perineum Care Knowledge Test will be redistributed and collected as a posttest upon completion of the training.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study
* Hhose mother tongue is Turkish,
* 18 years old and over
* Able to read and write

Exclusion Criteria:

* Who refused to participate in the study
* Native language is not Turkish
* Illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Palliative care patient relatives' perineum care information: First test | Just before training
  "Perineum Care Knowledge Test" is a test prepared by researchers in line with the literature and sent to an expert academician to ensure content validity. The Perineum Care Knowledge Test is a 3-likert-type questionnaire consisting of a total of 15 questions coded as true, false, I don't know. The minimum score to be obtained from the test is 0 and the maximum score is 15. A high score at the end of the evaluation indicates that the relatives of the patients have a high level of knowledge about perineal care, while a low score indicates a low level of knowledge.

SECONDARY OUTCOMES:
Perineal care information of palliative care patient relatives: Second test | Immediately after training
  "Perineum Care Knowledge Test" is a test prepared by researchers in line with the literature and sent to an expert academician to ensure content validity. The Perineum Care Knowledge Test is a 3-likert-type questionnaire consisting of a total of 15 questions coded as true, false, I don't know. The minimum score to be obtained from the test is 0 and the maximum score is 15. A high score at the end of the evaluation indicates that the relatives of the patients have a high level of knowledge about perineal care, while a low score indicates a low level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Nur Uzun, PhD, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department; Hümeyra Hançer Tok, PhD, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.